CLINICAL TRIAL: NCT06850974
Title: Foley Balloon for Cervical Preparation Before Dilation and Evacuation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Sierra Washington, MD, Clinical Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2023-00297; stony brook university (Other: stony brook university)
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Abortion, Second Trimester; Abortion, Medical
Keywords: second; trimester; abortion; surgical; balloon; Foley
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: single blind randomized controlled trial
Who Masked: Care Provider, Investigator
Masking Description: the providers performing the D&E is blinded to the cervical preparation type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Foley Balloon and misoprostol (Experimental): Patients in the Foley Balloon arm will have a Foley balloon catheter placed trans-cervically and also receive misoprostol per protocol
  Interventions: Device: Foley Balloon Catheter; Drug: Misoprostol
- Laminaria (Active Comparator): Patients in the Laminaria arm will have a Laminaria placed in the cervix and it will be left in situ per protocol
  Interventions: Device: Laminaria

INTERVENTIONS:
Device: Foley Balloon Catheter — 18 French Foley Balloon placed trans-cervically and inflated with 30-60ml of Normal Saline.
  Arms: Foley Balloon and misoprostol
Drug: Misoprostol — 400 mcg of buccal misoprostol sublingual
  Arms: Foley Balloon and misoprostol
Device: Laminaria — Laminaria will be placed in the cervix according to the following standard formula: Estimated gestational age -10 = number of 5mm laminaria.
  Arms: Laminaria

SUMMARY:
To evaluate the Foley Balloon technique for cervical preparation before second trimester surgical abortion between 16 and 21 weeks estimated gestational age in combination with misoprostol to prepare the cervix before dilation and evacuation (D&E) instead of osmotic dilators (Laminaria).

Specific Aim One: Assess definitively whether using a Foley Balloon and Misoprostol is non-inferior to osmotic dilators for cervical preparation before D&E.

Specific Aim Two: Evaluate patient satisfaction with the two methods of second trimester abortion.

Specific Aim Three: Evaluate provider satisfaction with the two methods of second trimester abortion.

DETAILED DESCRIPTION:
Termination of pregnancy was legalized in Mozambique in 2016 for any reason until 12 weeks, and up 16 weeks in cases of rape, and at any time for cases of fetal demise, severe fetal anomaly, or to protect a woman's physical or mental health. It is also legal up until 24 weeks in the case of a chronic infectious or degenerative disease. Termination of pregnancy can be accomplished either by induction of labor or by Dilation and Evacuation (D&E). Typically, D&E after 16 weeks is a two-day procedure. The first day is devoted to cervical preparation, where osmotic dilators are placed into the cervix and allowed to slowly soften and dilate the cervix. On the second day of the procedure the uterus is evacuated. Osmotic dilators are expensive and unavailable in most of Sub-Saharan Africa. An alternative strategy to cervical preparation has recently been developed by Dr. Yashica Robinson and has been described in a retrospective cohort study. This new technique involves using a Foley Catheter balloon (FB) inserted into the cervix to dilate the cervix over several hours with buccal misoprostol as an adjunct medication. After which, the procedure is completed using the dilation and evacuation procedure. However, Foley Balloon for cervical preparation before dilation and evacuation is still considered investigational. Both Foley Balloon and misoprostol are low cost and widely available in Africa and thus may be a safe and efficacious alternative to osmotic dilators. These two strategies of cervical preparation have never been directly compared in a prospective randomized clinical trial. This study aims to conduct a randomized controlled trial to evaluate the Foley Balloon for cervical preparation before D&E. Specifically, our objective is to evaluate the Foley Balloon technique for cervical preparation before second trimester surgical abortion between 16 and 21 weeks estimated gestational age. The investigators propose to conduct a randomized controlled non-inferiority trial to compare procedure difficulty, complication rates, provider satisfaction, and patient satisfaction with a novel technique to prove that the Foley Balloon and misoprostol method is safe, effective, and acceptable to providers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older presenting to Hospital Central de Maputo requiring abortion for any legal indication between 16-21 weeks gestation.
* Portuguese speaking

Exclusion Criteria:

* Less than age 18
* Incarcerated
* Chorioamnionitis
* Active heavy bleeding
* A known bleeding diathesis
* Hemodynamic instability
* > 2 cm dilation
* History of cervical cerclage
* Allergy to any study medications
* Eclampsia
* Glasgow Coma Score Less than 15

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients will be female confirmed pregnant patients
Enrollment: 102 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Total Procedure Time (TPT) | through completion of D&E, approximately 15-20 minutes
  Determine if Foley Balloon arm (misoprostol and foley balloon) is different to Laminaria arm (Laminaria only) in changing Total Procedure Time (TPT) of dilation and evacuation (D&E) procedure.

SECONDARY OUTCOMES:
D&E operative time (OT) | through completion of D&E, approximately 15-20 minutes
  Determine if Foley Balloon arm (misoprostol and foley balloon) is different to Laminaria arm (Laminaria only) in changing D&E operative time (OT) of dilation and evacuation (D&E) procedure.
Initial pre-operative cervical dilation | through completion of D&E, approximately 15-20 minutes
  Determine if Foley Balloon arm (misoprostol and foley balloon) is different to Laminaria arm (Laminaria only) in changing the initial pre-operative cervical dilation during the dilation and evacuation (D&E) procedure.
Potential Complications | through completion of the D&E, an average of 1-2 days
  Determine any potential same day complication rates between the foley balloon arm (foley balloon and misoprostol) versus the laminaria arm (laminaria only).
Visual Analogue Pain Scale | through completion of the D&E, an average of 1-2 days.
  Determine if Foley Balloon arm (misoprostol and foley balloon) is different to Laminaria arm (Laminaria only) in changing the pain rating before and after dilation and evacuation (D&E) procedure. Patient will complete a short survey, the Visual Analogue Pain Scale to rate their pain. The Minimum value of 0 and Maximum value of 10 where the higher value indicates more pain or worse outcome.
Provider Satisfaction Questionnaire | through study completion, an average of 1-2 days
  Providers will describe satisfaction by responding to questionnaire regarding cervical preparation.
Patient Satisfaction Questionnaire | through completion of the D&E, an average of 1-2 days
  Patients will describe satisfaction by responding to questionnaire regarding satisfaction with the cervical preparation procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Central De Maputo, Maputo, Cidade de Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
de-identifed patient database will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1/2026-1/2046
Access Criteria: Independent validated investigators, peer reviewed journal editors will be able to access the study protocol, the data analysis plan and the de-identified database should they wish to perform a meta- analysis.